CLINICAL TRIAL: NCT01436734
Title: Role of Aprotinin in Glucagon Degradation, Measurement by Radioimmunoactive Method (RIA) I125
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Mikkel Christensen, MD, University Hospital, Gentofte, Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-D-2009-0078
Record Dates: First submitted 2011-09-08; First posted 2011-09-20 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Hyperglucagonemia
MeSH Terms: interventions — Hig1 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GIP (Experimental)
  Interventions: Other: Fasting glycemia; Other: Hypoglycemia

INTERVENTIONS:
Other: Fasting glycemia — no intervention
Other: Hypoglycemia — Insulin induced hypoglycemia

SUMMARY:
The aim of the study was to investigate the role of the Trasylol in glucagon prevention in degradation using radioimmunoactive method with I125. Additionally different incubation time was introduced in human plasma samples after oral glucose stimulation, also in fasted and hypoglycemia blood samples from patients' type 2 diabetes. Since, the structure and the techniques for the glucagon measurement are well described nowadays.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians 18 years or older with Type 2 diabetes (WHO criteria)

Exclusion Criteria:

* HbA1c >9 %
* Liver disease (ALAT/ASAT >2 x upper normal limit)
* Diabetic nephropathy (s-creatinine >130 µM or albuminuria)
* Proliferative diabetic retinopathy (anamnestic)
* Severe arteriosclerosis or heart failure (NYHA group III og IV)
* Anemia
* treatment with medication not applicable to pause for 12 hours
* pregnancy or lactation
* Fasting plasma glucose >15 mM on screening day.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in plasma glucagon values measured with c-terminal specific "micro-protocol" RIA4305: 350µl of plasma (duplicate sample). | 120 min

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Christensen, MD, Principal Investigator — Gentofte Hospital
Locations (1):
- Gentofte Hospital, Hellerup, Denmark